CLINICAL TRIAL: NCT04589715
Title: Effect of Electroacupuncture on Symptoms of Female Pelvic Organ Prolapse(Level II - III )
Brief Title: Effect of Electroacupuncture on Symptoms of Female Pelvic Organ Prolapse(Level II - III)
Acronym: EAPOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Shaanxi Hospital of Traditional Chinese Medicine (Other); Hunan University of Traditional Chinese Medicine (Other); Lianyungang City Hospital of Traditional Chinese Medicine (Unknown); Jiangsu Second Hospital of Traditional Chinese Medicine (Unknown); Shenzhen Second People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Zhishun, Chief Physician, Dean of Acupuncture Department, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-249-KY-01
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Pelvic Organ Prolapse
Keywords: electroacupuncture; sham acupuncture; randomised controlled trial; Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: Patients who sign the informed consent form and are eligible for the study entry at week 0 will be randomized to one of the two groups: electroacupuncture group and sham electroacupuncture group. The two groups will be assessed in a paralleled manner, and patients in both groups will be treated for 24 times in 3 months(3 times weekly for 4 weeks, 2 times weekly for 4 weeks and once every week for 4 weeks) and followed up for 6 months after treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants, investigator and outcome assessor will be masked. The care provider cannot be masked, but will be different person from investigator and outcome assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electroacupuncture group (Experimental): patients will receive electroacupuncture at 3 acupoints(Bladder meridian of foot-taiyang 33 and 35#BL33 and BL35), and Spleen meridian of foot-taiyin 33(SP6)) 3 times/week for 4 weeks, then 3 times/week for 4 weeks, and then once/week for 4 weeks(24 times in total in 3 months), and be followed up for 6 months after treatment. Disposable acupuncture needles with size of 0.30 × 75 mm will be used at BL 33 and BL 35, and needles with size of 0.30 ×40 mm at SP 6. Standardized electroacupuncture apparatuses will be used, and the stimulation will last for 30 minutes with a continuous wave of 20 Hz, and a current intensity of 2 to 6.5 mA at BL33 and BL 35, and 1 to 3.5 mA at SP6.
  Interventions: Other: electroacupuncture
- sham electroacupuncture group (Sham Comparator): patient will receive sham electroacupuncture with the same frequency and amount as applied in the electroacupuncture group, as well as the follow-up period. Disposable acupuncture needles with size of 0.30 × 40 mm will be applied and penetrate the skin of patients for 2 to 3mm at sham acupoints to the 3 acupoints mentioned above. The stimulation will only last for 30-second with a very weak currency intensity and a continuous wave of 20 Hz.
  Interventions: Other: sham electroacupuncture

INTERVENTIONS:
Other: electroacupuncture — the same as described in experimental arm.
  Arms: electroacupuncture group
Other: sham electroacupuncture — the same as described in sham comparator.
  Arms: sham electroacupuncture group

SUMMARY:
The purpose of the study is to assess the efficacy and safety of electroacupuncture among women with pelvic organ prolapse(Level II - III), compared with sham electroacupuncture.

DETAILED DESCRIPTION:
After being informed about the study and potential risk, all patients giving written informed consent form will be undergo a 1-week screening period to determine eligibility for study entry. Eligible patients will be randomly assigned to one of the two groups 1) electroacupuncture group: electroacupuncture will be provided to patients at BL33, BL35 and SP6 for 3 time per week for the first 4 weeks, then twice a week for 4 weeks, and once a week for the last 4 weeks. There will be 24 times of treatment in total in 3 month; 2) sham electroacupuncture group: sham electroacupuncture will be provided to patients at sham acupoints to BL33, BL35 and SP6 with the same schedule as electroacupuncture group.The follow-up time for the two groups are 6 months after treatment. Primary and secondary outcome will be measured at 3, 6, and 9 months from the start of the treatment, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. female patients with pelvic organ prolapse at level 2-3 via POP-Q examination;
2. patients at the age of 35 years or older;
3. patients who have a sensation of bulging or protrusion from virginal area, with or without urinary, bowel, and sexual disorders;
4. patients who have a score of PFDI-20 > 24.
5. Patients who have signed informed consent form and are willing to participate the study voluntarily.

Patients will be included if all above 5 items are met.

Exclusion Criteria:

1. Patients who have cognitive disorders and cannot understand the content of questionnaires;
2. Patients who have severe heart, lung, brain, liver, kidney, hematopoietic system, and immune system diseases, or severe malnutrition;
3. Patients who have cancer or are at terminal stage of severe diseases;
4. Patients who need finger assistance for defecation, or have severe prolapse of rectum, sigmoid colon or small intestine;
5. Patients who have received(or are receiving) treatments for pelvic floor disorders , including pelvic organ prolapse, stress urinary incontinence, and etc in the past one month;
6. Patients who are receiving any treatment for other gynecological diseases;
7. Patients who have symptomatic urinary tract infection with urinary pain and urge, or have residual urine volume ≥ 100ml;
8. Patients who have diseases affecting the neurological function of pelvic organ, e.g. spinal cord injury, or peripheral nerve injury caused by surgery at lumbosacral area or pelvic floor .

Patients will be excluded if they meet any of the above criteria.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-10-31 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
the change from baseline on the score of the Pelvic Floor Distress Inventory-short form 20 (PFDI-20) | at baseline, and 3 months when the treatment is completed.
  Data will be collected via the the Pelvic Floor Distress Inventory-short form 20 (PFDI-20) . The questionnaire consists of three sections, pelvic organ prolapse distress inventory 6 (POPDI-6), colorectal-anal distress inventory 8 (CRADI-8), and urinary distress inventory 6 (UDI-6). Each section has 6-8 questions with 5 answers rated from 0-4 in each, and mean score of each section is the total score of this section divided by number of questions in this session. Then the sum of the mean scores of the three section timing 25 will come to the total score of the questionnaire(0-300). The higher the total score is, the severer the symptoms are.

SECONDARY OUTCOMES:
the change from baseline on the score of the Pelvic Floor Distress Inventory-short form 20 (PFDI-20) | 6 months and 9 months since the start of the treatment.
  Data will be collected via the Pelvic Floor Distress Inventory-short form 20 (PFDI-20) . The questionnaire consists of three sections, pelvic organ prolapse distress inventory 6 (POPDI-6), colorectal-anal distress inventory 8 (CRADI-8), and urinary distress inventory 6 (UDI-6). Each section has 6-8 questions with 5 answers rated from 0-4 in each, and mean score of each section is the total score of this section divided by number of questions in this session. Then the sum of the mean scores of the three section timing 25 will come to the total score of the questionnaire(0-300). The higher the total score is, the severer the symptoms are.
number of patients at different levels of pelvic organ prolapse quantitative examination(POP-Q) | at baseline, and 3 months when the treatment is completed.
  Pelvic organ prolapse quantitative examination(POP-Q) is a manual approach to measure the severity of female pelvic organ prolapse with five level from 0 to 4 . The POP-Q examination will be conducted by experienced gynecologists in each participating center. The higher the level is, the severer the symptoms are.
the change from baseline on the score of the Pelvic Floor Impact Questionnaire Short Form-7（PFIQ-7） | at baseline, 3 months, 6 months and 9 months since the start of the treatment.
  Data will be collected via the Pelvic Floor Impact Questionnaire Short Form-7（PFIQ-7) , which uses 7 questions to evaluate the impact of bladder, colorectal and virginal symptoms on daily life, respectively. For each type of symptoms, the answer to one question has four levels, no bother(0), mild bother(1), moderate bother(2), severe bother(3). The higher the total score is, the severer the quality of life is impacted.
the change from baseline in the validated Chinese version of International Consultation on Incontinence Questionnaire- Short Form(ICIQ-SF) scores | at baseline, 3 months, 6 months and 9 months since the start of the treatment.
  Data will be collected via International Consultation on Incontinence Questionnaire-Short Form(ICIQ-SF) questionnaire. The total score(0-21scores) is an accumulated scores from question 1 to 3. The higher the total score is, the severer the incontinence is.
the change from baseline on the score of pelvic organ prolapse/urinary incontinence sexual questionnaire-12(PISQ-12) | at baseline, 3 months, 6 months and 9 months since the start of the treatment.
  Data will be collected via pelvic organ prolapse/urinary incontinence sexual questionnaire-12(PISQ-12), which uses 10 questions to evaluate the impact of pelvic organ prolapse/urinary incontinence on sexual life for patients. The answer to each question has five levels, including always(4), often(3), sometimes(2), rarely(1), never(0). The higher the total score is, the severer the impact of pelvic organ prolapse/incontinence to sexual life is.
score of the patient global index of improvement (PGI-I) | at baseline, 3 months, and 9 months since the start of the treatment.
  Data will be collected via the Patient Global Index of Improvement (PGI-I) to evaluate the overall treatment effect from patient's perspective. Patient will be asked about their feelings on change of symptoms after treatment. The change can be rated in 7 levels, including major improvement, moderate improvement, mild improvement, no improvement, mild worsening, moderate worsening, and major worsening.
patients' expectation to the effect of treatment | at baseline, and 3 months when the treatment is completed.
  patients will be asked about their expected effect of the treatment via question: In your expectation, how is your symptoms like in three month. Five choices will be provided 1) much better; 2) slightly better; 3) I don't know; 4)no change; 5) worse.
incidence rate of any adverse events | 3 months, 6 months and 9 months since the start of the treatment.
  numbers and types of any adverse event associated either with or without acupuncture will be documented as soon as it is reported in any centers. The incidence rate of adverse event will be analyzed and reported.
blinding assessment | in 12th week after any acupuncture treatment
  patients will be asked whether they received electroacupuncture or sham acupuncture to assess the effect of blinding.

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, PhD,MD, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: No
We cannot share IPD under current regulation of Human Genetic Resources Management in China.

REFERENCES:
- [Derived] Chen H, Liu X, Yan Y, Shi H, Liu Z. Effect of electroacupuncture on symptoms of female pelvic organ prolapse (stage II-III) (EAPOP study): protocol of a randomised controlled trial. BMJ Open. 2022 Jun 6;12(6):e051249. doi: 10.1136/bmjopen-2021-051249. PMID 35667733